CLINICAL TRIAL: NCT03319836
Title: Meeting Protein Targets in Critically Ill Patients: A Retrospective Analysis
Brief Title: Meeting Protein Targets in Critically Ill Patients
Acronym: PROTARGET
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 16.02.CA.HCN
Record Dates: First submitted 2017-09-19; First posted 2017-10-24 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Critical Illness; Dietary Modification
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-very high protein enteral nutrition: 20 enterally fed critically ill adult patients prior to the introduction of a very high protein enteral nutrition formula [2015].
- Post-very high protein enteral nutrition: 20 enterally fed critically ill adult patients post the introduction of a very high protein enteral nutrition formula [2016].

SUMMARY:
This is a retrospective study of protein and energy intake in enterally fed critically ill adult patients before and after the introduction of a very high protein enteral nutrition formula in a single center medical/surgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age, mechanically ventilated
* Received enteral nutrition for a minimum of five days during the first week of ICU admission

Exclusion Criteria:

* Received parenteral nutrition during first week of ICU admission
* Acute renal failure not dialyzed
* Hepatic encephalopathy grade 3 or 4
* Intentional underfeeding/trophic feeding - including refeeding syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult medical/surgical ICU patients that received enteral nutrition with or without a very high protein enteral nutrition formula.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Daily total protein intake | Daily up to 7 days of ICU stay
  Daily total protein intake and percent prescribed protein needs met during first week of ICU admission.

SECONDARY OUTCOMES:
Daily caloric intake - Total Calories | Daily up to 7 days of ICU stay
  Total calories aggregate from all sources
Daily caloric intake - kcal/kg | Daily up to 7 days of ICU stay
  Total volume consumed and weight will be used to measure kcal/kg
Daily caloric intake from enteral nutrition | Daily up to 7 days of ICU stay
  Daily caloric intake from enteral nutrition, and medications (i.e. Propofol)
Percentage of prescribed calorie needs met | Daily up to 7 days of ICU stay
  Percentage of prescribed calorie needs met
Feeding interruptions | Daily up to 7 days of ICU stay
  Feeding interruptions; and reason for interruption, if recorded in electronic medical record/nursing flow sheets
Use of inotropes/vasopressors (highest daily dose prescribed) | Daily up to 7 days of ICU stay
  Use of inotropes/vasopressors will be documented as a Yes/No.
Feeding tolerance | Daily up to 7 days of ICU stay
  Feeding tolerance as recorded by clinicians in electronic medical record/nursing flow sheets [gastrointestinal side effects observed and documented: vomiting, elevated Gastric Residual Volumes (>200 mL), aspiration, pneumonia, diarrhea (Bristol stool chart definition and ≥ 3 liquid stools/day)]

CONTACTS AND LOCATIONS:
Overall Officials: Michele ApSimon, Principal Investigator — Hamilton Health Sciences Centre
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No